CLINICAL TRIAL: NCT03121638
Title: An Open Label, Active Controlled, Parallel Group Phase I Clinical Trial to Assess the Safety, Tolerability and Immunogenicity of NBP608 in Healthy Adult Volunteers
Brief Title: Safety Study of NBP608 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NBP608_VZ_I_2012
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Varicella Zoster; Immunization; Infection
Keywords: Varicella Vaccine; Herpes Zoster Vaccine
MeSH Terms: conditions — Infections | interventions — Chickenpox Vaccine; Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- VARIVAX (Active Comparator): Single dose 0.5mL of Varivax by subcutaneous injection into the outer aspect of the upper arm
  Interventions: Biological: VARIVAX
- ZOSTAVAX (Active Comparator): Single dose 0.65mL of Zostavax by subcutaneous injection into the outer aspect of the upper arm
  Interventions: Biological: ZOSTAVAX
- NBP6081 (Experimental): Single dose 0.5mL of low potency of NBP608 by subcutaneous injection into the outer aspect of the upper arm
  Interventions: Biological: NBP6081
- NBP6082 (Experimental): Single dose 0.5mL of middle potency of NBP608 by subcutaneous injection into the outer aspect of the upper arm
  Interventions: Biological: NBP6082
- NBP6083 (Experimental): Single dose 0.5mL of high potency of NBP608 by subcutaneous injection into the outer aspect of the upper arm
  Interventions: Biological: NBP6083

INTERVENTIONS:
Biological: VARIVAX — Preparation of Oka/Merck strain of live, attenuated varicella zoster virus
  Arms: VARIVAX
Biological: ZOSTAVAX — Preparation of Oka/Merck strain of live, attenuated varicella zoster virus
  Arms: ZOSTAVAX
Biological: NBP6081 — Preparation of Oka/SK strain of live, attenuated varicella zoster virus
  Arms: NBP6081
Biological: NBP6082 — Preparation of Oka/SK strain of live, attenuated varicella zoster virus
  Arms: NBP6082
Biological: NBP6083 — Preparation of Oka/SK strain of live, attenuated varicella zoster virus
  Arms: NBP6083

SUMMARY:
* Indication: Protection against varicella and herpes zoster
* Study Objectives

  * Primary: Safety and tolerability assessment after single dose administration of NBP608
  * Secondary: immunogenicity assessment after single dose administration of NBP608

DETAILED DESCRIPTION:
This is a single-center, open label, active controlled, dose-escalation, parallel group study to assess the safety, tolerability and immunogenicity of NBP608 in healthy adult volunteers. Total of 150 healthy subjects aged 20 and over are enrolled, and each subject is administered with single dose of vaccine which is sequentially assigned to active group 1, 2 and study group 1~3 in 1:1:1:1:1 ratio(30 subjects are enrolled at each groups) .

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 20 and over
* Availability to volunteer for the entire study duration and willing to adhere to all protocol requirements
* Female subjects of post-menopausal (amenorrhea for 24 months) whose pregnancy tests was found negative at screening visit
* Subjects of seropositive for Varicella-Zoster virus at screening visit

Exclusion Criteria:

* Patients with herpes zoster
* Subjects with a history of vaccination for herpes zoster
* Pregnant or lactating women
* Participants in another clinical study within 4 weeks before vaccination in this study, etc.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Incidence Rate of Adverse Event | 42days after Investigation Product Vaccination

SECONDARY OUTCOMES:
Varicella Zoster Virus Antibody Titer Measured by FAMA(Fluorescent Antibody to Membrane Antigen) | 42days after Investigation Product Vaccination
Varicella Zoster Virus Antibody Titer Measured by gpELISA(Glycoprotein Enzyme-Linked Immunosorbent Assay) | 42days after Investigation Product Vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Hee-jin Cheong, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No